CLINICAL TRIAL: NCT00146354
Title: The Effects of a Results Management System on Physician Awareness of Post-Discharge Laboratory and Radiology Results
Brief Title: The Effects of a Results Management System on Physician Awareness of Post-Discharge Test Results
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Risk Management Foundation (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: 2003P000551
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2005-08

CONDITIONS: Healthy; Medical Record Systems, Computerized
Keywords: Electronic Medical Record; Electronic Results Tracking; Patient Safety; Post-Discharge Test Results

INTERVENTIONS:
Behavioral: Hospitalists Results Manager

SUMMARY:
This project aims to define the problem of results that return after patient discharge and to study the implementation of an Electronic Medical Record (EMR)-based system for tracking these results.

DETAILED DESCRIPTION:
The transfer of care at hospital discharge is complex and requires the transmission of large amounts of data between inpatient physicians (hospitalists) and outpatient physicians (PCPs), including information about pending tests. Frequently, laboratory and radiology tests are not finalized until after a patient is discharged, and when the responsibility for these pending results is not clearly defined, they can be missed. Our project aims to define the problem of these post-discharge results and to study the implementation of an EMR-based system (Hospitalist Results Manager, HRM) for tracking these results on the hospitalist services at Brigham and Women's Hospital (BWH) and Massachusetts General Hospital (MGH). The project consists of two phases: a cross-sectional study before intervention to define the epidemiology of post-discharge results, and a randomized trial of HRM to determine its effect on physician awareness of these results.

ELIGIBILITY:
Inclusion Criteria:

* Admitted under enrolled study Attendings at the two study locations
* Patient had test result finalized after discharge and prior to subsequent admission

Exclusion Criteria:

* Test result noted in discharge summary
* Test result not clinically actionable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tejal K Gandhi, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts